CLINICAL TRIAL: NCT06923176
Title: Effect of Biejia-Ruangan Compound on Survival Rate and Recurrence Rate of Hepatocellular Carcinoma After Radical Treatment
Acronym: BRCSRRRHCCART
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhiyun Yang (Other)
Responsible Party: Sponsor-Investigator, Zhiyun Yang, Vice President of Beijing Ditan Hospital Affiliated to Capital Medical University, Beijing Ditan Hospital
Organization: Beijing Ditan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJDHYZYBRC
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): Conventional treatment
  Interventions: Other: Routine medical care
- Treatment group (Experimental): Conventional treatment plus Biejia-Ruangan compound
  Interventions: Drug: Biejia-Ruangan compound; Other: Routine medical care

INTERVENTIONS:
Drug: Biejia-Ruangan compound — Biejia-Ruangan compound have the functions of softening hardness, dispersing lumps, removing blood stasis and detoxifying, and nourishing qi and blood. Used for chronic hepatitis B liver fibrosis, as well as early liver cirrhosis characterized by blood stasis obstructing collaterals, qi and blood deficiency with incomplete heat toxicity.
  Arms: Treatment group
Other: Routine medical care — Routine medical care

SUMMARY:
This study plans to enroll 704 patients with a history of chronic hepatitis B who have undergone radical treatment for hepatocellular carcinoma. The subjects were divided into a control group (conventional treatment group) and a combination therapy group (conventional treatment plus Biejia-Ruangan compound) according to the doctor's clinical diagnosis and treatment and the subjects' wishes in a ratio of 1:2. The subjects in the combination therapy group were treated with Biejia-Ruangan compound for 72 weeks, followed by 168 weeks of follow-up, for a total study period of 240 weeks.

By analyzing the 1-, 2-, 3-, and 5-year recurrence-free, overall survival rate/survival time, adverse reactions, etc., the clinical effect of Biejia-Ruangan compound in reducing the risk of recurrence in patients with hepatocellular carcinoma after receiving radical treatment was comprehensively evaluated, and its scientific value and practical application prospects as a potential treatment method were explored.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-75 years old (including 18 and 75 years old), regardless of gender.
* Individuals with chronic hepatitis B liver fibrosis or cirrhosis.
* According to the "Diagnosis and Treatment Guidelines for Primary Liver Cancer" (2024 edition) liver cancer diagnosis roadmap, the first clinical diagnosis is Hepatocellular carcinoma(HCC).
* The staging of liver cancer is CNLC stage Ia - IIa.
* Radical treatment has been completed, with surgical resection or local ablation.
* 8-12 weeks after radical surgery, imaging and serological evaluations showed no residual cancerous lesions and no new cancerous lesions were found.
* Child Pugh score A/B.
* Voluntarily joining the group, able to understand and sign an informed consent form.

Exclusion Criteria:

* Pregnant and lactating women;
* Prior to radical liver cancer surgery, the patient had received radiation, chemotherapy, molecular targeting, immunotherapy, and other anti-tumor treatments;
* Receive other anti-tumor Chinese medicine (including traditional Chinese patent medicines and simple preparations or Chinese herbal medicine);
* Individuals with mental illnesses, especially those with a history of depression, anxiety, mania, schizophrenia, or a family history of mental illness (especially those with a history of depression or tendencies towards depression);
* Combination of hepatitis A, C, D, E, and/or current HIV infections;
* Kidney diseases: acute and chronic nephritis, renal insufficiency, nephrotic syndrome, etc., or screening with blood creatinine>2.0 × ULN;
* Autoimmune diseases, including psoriasis, systemic lupus erythematosus, autoimmune liver disease, etc;
* Patients who experience upper gastrointestinal bleeding within the first 3 months (including the screening period) prior to screening;
* Individuals with a serious history of heart disease, especially those with unstable or poorly controlled heart disease within the past 6 months;
* Individuals who plan to receive organ transplantation or have already undergone organ transplantation;
* Those who are allergic to Compound Biejia Ruangan Tablets, nucleoside (acid) analogues, or drug excipients, or who meet any contraindications in the experimental drug instructions;
* Have used other anti fibrotic drugs within the first 6 months of enrollment, such as Fuzheng Huayu, Anluo Huaxian, and Ganshuang Granules.
* Other situations where the participant has participated in other intervention trials within the previous month or where the researcher deems it unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Estimated)
Dates: Start 2025-04-19 (Estimated); Primary Completion 2031-04-30 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 96 weeks

SECONDARY OUTCOMES:
Overall survival rate | 96 weeks
quality of life (QOL) questionnaire | 96 weeks
  The questionnaire includes appetite, sleep, fatigue, pain, etc.